CLINICAL TRIAL: NCT06027359
Title: The Effect of therapeutıc Game on nursıng ınıtıatıves and Fears of medıcal materıals ın Preschool chıldren
Brief Title: The Effect of therapeutıc Game on Preschool chıldren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Filiz KARACA DEVELİ, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: AdnanMU-ÇSHH-FKD-01
Record Dates: First submitted 2023-08-24; First posted 2023-09-07 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Fear; Nurse; Hospital
Keywords: Fear, hospital, nurse, play therapy, preschool
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Therapeutic game to reduce fear of hospital and ambulance (Experimental): therapeutic play was applied to 5 groups every day of the week and was completed in 4 weeks.
  Interventions: Other: Therapeutic play hospital fear and nursing interventions
- Therapeutic game to reduce fear of injectors and eye drops (Experimental): therapeutic play was applied to 5 groups every day of the week and was completed in 4 weeks.
  Interventions: Other: Therapeutic play hospital fear and nursing interventions
- Therapeutic play to reduce fear of intrauterine and serum (Experimental): therapeutic play was applied to 5 groups every day of the week and was completed in 4 weeks.
  Interventions: Other: Therapeutic play hospital fear and nursing interventions
- Therapeutic play to reduce fear of EKG and EMG (Experimental): therapeutic play was applied to 5 groups every day of the week and was completed in 4 weeks.
  Interventions: Other: Therapeutic play hospital fear and nursing interventions

INTERVENTIONS:
Other: Therapeutic play hospital fear and nursing interventions — Children assigned to the study group will be divided into 5 groups, with a maximum of 8 children. The researcher will perform a therapeutic play activity with each group consisting of maximum 8 children one day of the week in the room and time determined by the school. Each activity will last an average of 30 minutes. Therapeutic play activities will be completed in 4 weeks.
  * Therapeutic play activities will not be performed with the children in the control group.
  * One week after the completion of the therapeutic play intervention, the researcher will re-fill the Child Nursing Interventions and Fear of Materials Scale-uncommon materials sub-dimension face-to-face with the children in the study and control groups.

SUMMARY:
In processes such as illness, hospital, medical procedures, and nursing interventions, the fears experienced by children should be reduced before the procedure. It may be more effective to give interventions to reduce children's fears in a school setting rather than in a complex environment such as a hospital. In this context, there is a need for experimental studies that reveal the effect of therapeutic play on nursing interventions and fear of medical materials in preschool children.

DETAILED DESCRIPTION:
Entrance: In processes such as illness, hospital, medical procedures, and nursing interventions, the fears experienced by children should be reduced before the procedure. It may be more effective to give interventions to reduce children's fears in a school setting rather than in a complex environment such as a hospital. In this context, there is a need for experimental studies that reveal the effect of therapeutic play on nursing interventions and fear of medical materials in preschool children.

Aim: This study was planned to determine the effect of therapeutic play on nursing interventions and fear of medical materials in preschool children.

Method/ Data Collection Techniques:This research was planned as a quasi-experimental study with pretest-posttest and control group. The universe of the research will consist of 170 children studying in pre-school classes at the Chamber of Commerce Primary School located in the city center of Aydın. The sample size of the study was calculated using G*power analysis and it was found that a total of 70 children (study: 35 children, control: 35 children). However, considering the losses from the research and the possibility of children filling in the questionnaires incomplete or incorrectly, the number of children was increased by 10% and it was planned to complete the study with 80 (study: 40 children, control: 40 children) children. It is planned to collect the data between March 1 and June 1, 2023. The child to be included in the study and their parents will be informed about the study, verbal consent will be obtained from the children and written consent will be obtained from the parents. After obtaining parental consent about the study, the parents of the children in both the study and control groups will have to fill in the "Introductory Information Form" and the children will fill in the "Scale of Fear of Nursing Interventions and Used Materials in Children" before the therapeutic play. The therapeutic game content to be applied to the study group consists of four sessions organized by considering nursing interventions and materials used in the hospital. In each session, various game activities will be held with different materials. Therapeutic play activity will not be planned for the children in the control group. One week after the therapeutic play activities are completed, the children will have to fill out the "Scale of Fear Against Nursing Interventions and Used Materials in Children".

The data obtained in the research will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Homogeneity of descriptive features between groups will be tested by chi-square analysis. The Kolmogorov Smirnov Test will be used to determine whether the research data are normally distributed. In the analysis of study data, descriptive statistics, if the data show normal distribution, independent group-t-test and changes within the group repeated measurements Anova test; If it does not have a normal distribution, Mann Whitney-U test and Wilcoxon signed-rank test will be used.

Expected Results: Thanks to the results obtained from this study, it is expected that the familiarity of children with nursing interventions and materials with the therapeutic play method in their own environment such as school will help them experience less fear and adapt easily during a possible hospital experience in the future.

ELIGIBILITY:
Inclusion Criteria:

Child's:

* Between 60 months and 71 months (children over 71 months are educated in the first grade of primary education).
* Having pre-school education
* Absence of any mental and/or physical health problems that would prevent communication belonging to the parent. Belonging to the parent;
* Literacy of the parents

Exclusion Criteria:

The child has any phobia or is receiving treatment for this issue.

Ages: 60 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Nursing interventions and fear of materials used in children scale | baseline and week 4
  I am not afraid (1) I am extremely afraid (5). As the score increases, fear increases.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz KARACA DEVELİ, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Filiz KARACA DEVELİ, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No